CLINICAL TRIAL: NCT06034353
Title: Impact of Pharmacist-led Cognitive Behavioral Intervention on Adherence and Quality of Life of Epileptic Patients
Acronym: COGNIPHARM-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Matti Ullah, Assistant Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NA0823
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy
Keywords: Cognitive behavioral therapy; Pharmacist; Medication Adherence; Quality of life
MeSH Terms: conditions — Epilepsy; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be entertained as part of their regular appointment for prescription filling without any information of which group they are assigned in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic group (Active Comparator): Lifestyle Modifications: General education about healthy life style and diet. Education : general awareness about disease and medication Pill Planner: Pill planner will be provided to keep them adherent to their medication Counselling: Counsel the patients about there medication dosage, frequency and appropriate time.
  Interventions: Behavioral: Pharmacist-led Cognitive Behavioral therapy
- Advanced (Experimental): Lifestyle Modifications: Specific education on keto-diet, yoga and meditation Education : Specific disease education targeting medication adverse drug reaction (ADR), seizure chart management Pill Planner: Pill planner will also be provided to this group Counselling: Cognitive Behavioral therapy will be provided
  Interventions: Behavioral: Pharmacist-led Cognitive Behavioral therapy

INTERVENTIONS:
Behavioral: Pharmacist-led Cognitive Behavioral therapy — Pharmacist-led Cognitive Behavioral therapy is patient centered approach that focus both physical and emotional aspect of health is provided. It is focused to identify negative and change negative thought pattern and behavior to improve mental and physical well being.Incorporation education about healthy meal choices, relaxation techniques, self management strategies,to improve education about potential adverse effect, how to recognize and on followup calls how to adjust medication doses along with this is provided.

SUMMARY:
The purpose of this interventional study is to assess the impact of pharmacist-led cognitive behavioral intervention in epileptic patients. The main questions are:

1. If pharmacist-led cognitive behavioral therapy can help in improving patient medication adherence?
2. How will the cognitive behavioral therapy impact the quality of life of the patients?

Participants of this study will be provided basic or advanced level counselling and educational material as part of their routine pharmacy visit.

Researchers will compare the two groups (Basic and advanced) to see which of the two groups are better in term of medication adherence and quality of life.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether incorporation of pharmacist-led cognitive behavioral therapy (CBT) to the treatment of epileptic patients can result in better adherence to anti epileptic drugs. In order to manage epilepsy effectively, medication adherence is essential. Missed doses or irregular drug use can increase the frequency of seizures and reduce the effectiveness of treatment. In order to improve medicine adherence rates, the study will examine if cognitive behavioral therapy (CBT) therapies can have a favorable effect on patients' motivation, coping techniques, Medication beliefs, reduction in adverse drug reaction (ADRs), Seizures frequency and medication related problems (MRPs) other than adverse drug reaction (ADRs) and overall quality of life of epileptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis.
* Patients treated for epilepsy with at least one anti epileptic drug, subjects willing to participate in the study with or without other severe co-morbidities were included in the study.

Exclusion Criteria:

* Pregnant female patients.
* Patients who provide incomplete information
* Patients with any terminal disease e.g., end stage renal disease
* Patients not willing to participate were excluded from the study.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 3 months
  Adherence will be assessed using (Medication Adherence Reporting Scale) MARS-10.
  This scale describes three-dimension, Medication adherence behavior (1-4), attitude towards taking medication (5-8), negative side effects and attitudes to psychotropic medication (9-10). Each question has Yes and No response, a response consistent with adherence is coded as 1 and with non-adherence coded as 0. Higher the score higher will be the adherence. Adherence <6 is poor adherence, and >8 is high adherence.
Quality of life of Epileptic patients | 3 months
  Patient's quality of life will be assessed using Quality of life for epilepsy scale(QOLIE-31). QOLIE-31(Quality of life in epilepsy) used for quality-of-life assessment which assess the patient's life's quality level along using anti-epileptic drug (AED) therapy through close ended questions with a score. The score can range from 0-100, with 100 representing the best quality of life.

SECONDARY OUTCOMES:
Incidence of Drug-Drug Interactions | 3 months
  Drug interactions among epileptic and non-epileptic drug will be assessed using standard website (update-Lexicomp) It is used to access the reduction in no. of drug drug interaction after pharmacist intervation in both basic and advance groups.
Incidence of Adverse reactions | 3 months
  Adverse reactions of all anti-epileptic drug will be noted while assessing a patient.
  It is used to access the reduction in frequency of Adverse drug reaction after pharmacist intervation in both basic and advance groups.
Rate of seizures per week | 3 months
  While assessing patient no. of seizures per week is asked and noted by the pharmacist. After intervening both basic and advance group impact of intervation is accessed for no. of seizures in the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Ullah, PhD, Study Director — Hamdard University Islamabad Campus; Iqra Farooq, MPhil, Principal Investigator — Shifa International Hospital; Muhammad Shafiq, BS. (Hons.), Study Chair — Subhan Medical Trust; Emmama Jamil, MPhil, Study Chair — Hamdard University Islamabad Campus
Locations (1):
- Shifa International Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Sharing patient data will depend on the patient's consent. If the patient doesn't allow to share data with others, we will not be able to share individual data.